CLINICAL TRIAL: NCT04983420
Title: Effects of Different Polyphenol-containing Beverages on the Immune System and on Muscular Growth Factors - a Pilot Study
Brief Title: Effects of Different Polyphenol-containing Beverages on the Immune System and on Muscular Growth Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Polyphenol
Record Dates: First submitted 2021-05-06; First posted 2021-07-30 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Food Sensitivity
MeSH Terms: conditions — Food Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- non-alcoholic Pilsner (Experimental): 1 L non-alcoholic Pilsner per day for 2 weeks
  Interventions: Other: non-alcoholic Pilsner
- non-alcoholic wheat beer (Experimental): 1 L non-alcoholic wheat beer per day for 2 weeks
  Interventions: Other: non-alcoholic wheat beer
- apple spritzer (Active Comparator): 1 L apple spritzer per day for 2 weeks
  Interventions: Other: apple spritzer
- lemonade (Placebo Comparator): 1 L lemonade per day for 2 weeks
  Interventions: Other: lemonade

INTERVENTIONS:
Other: non-alcoholic Pilsner — intake of 1 L non-alcoholic Pilsner per day for 2 weeks
  Arms: non-alcoholic Pilsner
Other: non-alcoholic wheat beer — intake of 1 L non-alcoholic wheat beer per day for 2 weeks
  Arms: non-alcoholic wheat beer
Other: apple spritzer — intake of 1 L apple spritzer per day for 2 weeks
  Arms: apple spritzer
Other: lemonade — intake of 1 L lemonade per day for 2 weeks
  Arms: lemonade

SUMMARY:
In this research project, the effect of different polyphenol-containing beverages with varying alcohol content of < 0.4 vol% on immune function as well as muscular growth factors will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 20 - 60 years
* Written informed consent

Exclusion Criteria:

* severe gastrointestinal disease or known malabsorption
* use of proton pump inhibitors
* malignancies
* rheumatoid diseases
* metabolic syndrome
* acute or chronic infections or inflammatory diseases
* use of medications or supplements to interfere with immune function
* alcohol and/or drug abuse or addiction
* dependent relationship with the project manager or his or her employees
* pregnancy or breastfeeding
* chronic illness or regular use of medication (except hormonal contraception)
* smoker

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
white blood cells | before beverage intake
  white blood cell count
white blood cells | 60 minutes after intake
  white blood cell count
white blood cells | 120 minutes after intake
  white blood cell count
inflammatory markers in the blood | before beverage intake
  IL-6, TNF- α, hs-CRP
inflammatory markers in the blood | 60 minutes after intake
  IL-6, TNF- α, hs-CRP
inflammatory markers in the blood | 120 minutes after intake
  IL-6, TNF- α, hs-CRP
blood alcohol | before beverage intake
  blood alcohol level
blood alcohol | 60 minutes after intake
  blood alcohol level
blood alcohol | 120 minutes after intake
  blood alcohol level
white blood cells | after 14 days of daily intake
  white blood cell count
inflammatory markers in the blood | after 14 days of daily intake
  IL-6, TNF- α, hs-CRP
blood alcohol | after 14 days of daily intake
  blood alcohol level
polyphenol in the urine | before beverage intake
  polyphenol level in the urine
polyphenol in the urine | 120 minutes after intake
  polyphenol level in the urine
polyphenol in the urine | after 14 days of daily intake
  polyphenol level in the urine

SECONDARY OUTCOMES:
dietary habit | before beverage intake and day 12-14 of beverage intake
  3 day food diary
dietary habit | day 12-14 of beverage intake
  3 day food diary
physical activity | before beverage intake
  Global Physical Activity Questionnaire (allows to calculate metabolic equivalents to express the intensity of physical activities
physical activity | day 14 of beverage intake
  Global Physical Activity Questionnaire (allows to calculate metabolic equivalents to express the intensity of physical activities

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Scherr, Prof, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No